CLINICAL TRIAL: NCT02020733
Title: Evaluation of Pain During Hysterosalpingography With The Use Of Balloon Catheter Versus Metal Cannula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sadiman Kiykac Altinbas (Other)
Responsible Party: Sponsor-Investigator, Sadiman Kiykac Altinbas, M. D., Etlik Zubeyde Hanim Womens' Health and Teaching Hospital
Organization: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20.12.13/160
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Pain During Hysterosalpingography
Keywords: Hysterosalpingography; balloon catheter; metal cannula; pain assessment

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- balloon catheter (Other)
  Interventions: Device: Balloon catheter
- metal cannula (Other)
  Interventions: Device: metal cannula

INTERVENTIONS:
Device: Balloon catheter
  Arms: balloon catheter
Device: metal cannula
  Arms: metal cannula

SUMMARY:
The aim of this study is to compare the metal cannula routinely used in our clinical practice with intrauterine hysterosalpingography catheter as a probable alternative device in a prospective, single-blinded, randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18-47 years,
* applying for basic infertility evaluation to the Reproductive Endocrinology unit

Exclusion Criteria:

* The patients with a known hypersensitivity to iodine or radio-opaque contrast dye,
* vaginal bleeding,
* genital malignancy and
* any sign of pelvic inflammatory disease (PID) were excluded

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 194 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
the degree of pain experienced during the procedure | 1 hour after the procedure
  The primary outcome was the degree of pain experienced during the procedure, pain was evaluated with the Wong Baker Faces Pain Rating Scale (WBS), which ranked the pain from 0 to 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik Zubeyde Hanim Women's Health Teaching and Research Hospital, Ankara, Turkey (Türkiye)